CLINICAL TRIAL: NCT07359066
Title: An Open-label, First-in-Human, Dose-Escalation and Dose-Expansion Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of SPR1020 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai SciBrunch Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPR1020-S-001
Record Dates: First submitted 2025-12-16; First posted 2026-01-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors; PARP Inhibitor
Keywords: SPR1020

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 25mg/day (Experimental)
  Interventions: Drug: SRP1020
- 50mg/day (Experimental)
  Interventions: Drug: SRP1020
- 100mg/day (Experimental)
  Interventions: Drug: SRP1020
- 150mg/day (Experimental)
  Interventions: Drug: SRP1020
- 200mg/day (Experimental)
  Interventions: Drug: SRP1020
- 250mg/day (Experimental)
  Interventions: Drug: SRP1020

INTERVENTIONS:
Drug: SRP1020 — SPR1020 is administered orally. The dosing frequency is once daily (QD). Each treatment cycle is 21 days.

SUMMARY:
This study is a multicenter, open-label study designed to evaluate SPR1020 in adult patients with advanced solid tumors. The study aims to characterize the safety, tolerability, pharmacokinetic (PK) profile, and preliminary antitumor activity of SPR1020 monotherapy in this population.

The study consists of two parts: Phase I component (dose escalation and backfill) and Phase II component (dose expansion). The primary objectives of the Phase I part are to investigate the safety, tolerability, and PK profile of SPR1020 and to determine the Recommended Phase II Dose (RP2D) and/or the Maximum Tolerated Dose (MTD), if attainable. The Phase II part will be initiated once the RP2D and/or MTD is established in the Phase I part.

As a new-generation, highly selective PARP1 inhibitor, SPR1020 demonstrates a competitive clinical benefit-risk profile, combining potential intracranial activity with a differentiated safety profile. By leveraging a "synthetic lethality" mechanism, SPR1020 is expected to demonstrate significant efficacy against tumors harboring BRCA mutations or homologous recombination repair (HRR) pathway gene alterations (e.g., breast cancer, prostate cancer). Owing to its high selectivity for PARP1 over PARP2, SPR1020 may circumvent the hematological toxicities associated with PARP2 inhibition by first-generation pan-PARP inhibitors (e.g., olaparib), potentially resulting in an improved safety profile. This enhanced safety may provide greater flexibility for use in combination therapies. Furthermore, SPR1020's ability to penetrate the blood-brain barrier could offer a new treatment option for patients with advanced disease and brain metastases, addressing a high unmet medical need in this population with limited therapeutic choices. Preclinical data support this differentiated profile in terms of both efficacy and toxicity.

Hypothesis: SPR1020 represents a novel anticancer therapeutic with the potential for enhanced efficacy and an improved safety profile. The overall assessment indicates that its clinical benefits outweigh the potential risks.

This study has been approved by the IEC and adheres to the principles of the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjets ≥ 18 years old.
2. Phase I Dose-Escalation Part: Patients with histologically or cytologically confirmed, surgically unresectable, locally advanced or metastatic malignant solid tumors, who have experienced failure of standard therapy, or for whom no standard therapy exists, or who are intolerant to standard therapy. (Priority will be given to enrolling patients with breast, ovarian, prostate, or pancreatic cancer harboring homologous recombination deficiency (HRD)-related gene mutations such as BRCA1/2, PALB2, RAD51C/D).

Phase I Dose Backfill Portion: Patients with HER2-negative breast cancer (BC), advanced epithelial ovarian cancer (OC)/fallopian tube cancer (FTC)/primary peritoneal cancer (PPC), or castration-resistant prostate cancer (CRPC), who have a documented pathogenic or likely pathogenic BRCA mutation (BRCAm, germline or somatic) as detected by a local or central laboratory, and who have experienced failure of at least one prior line of standard anticancer therapy (refer to the protocol section for the Phase II dose expansion for specific standard therapy requirements); Or patients with other tumor types harboring homologous recombination deficiency (HRD) related gene mutations (including but not limited to esophageal cancer, small cell lung cancer, or pancreatic cancer) who have experienced failure of at least one prior line of standard therapy.

Phase II Dose Expansion Study: Allows prior treatment with a pan-PARP inhibitor (no more than 1 type). Specific requirements for each cohort are as follows:

Cohort 1: Breast Cancer (BC):

1. Histologically or cytologically confirmed HER2-negative (HR+/HER2- or triple-negative) advanced or metastatic breast cancer.
2. Presence of a predicted loss-of-function BRCA1/2 mutation in germline or tumor tissue.
3. Received at least > 1 line of systemic therapy for advanced disease (must have received at least one line of chemotherapy; if HR+, must have received endocrine therapy), with recent radiological confirmation of disease progression.

Cohort 2: Ovarian Cancer (OC):

1. Histologically confirmed high-grade serous or endometrioid ovarian cancer, fallopian tube cancer, or primary peritoneal cancer.
2. Presence of a predicted loss-of-function BRCA1/2 mutation in germline or tumor tissue.
3. Received at least > 1 line of systemic therapy for advanced disease (must have received at least one platinum-based chemotherapy regimen for advanced disease), with recent radiological confirmation of disease progression.
4. Subjects must have a response duration of ≥ 6 months after the last platinum-based chemotherapy (platinum-sensitive population).

Cohort 3: Prostate Cancer (PC):

1. Histologically or cytologically confirmed prostatic adenocarcinoma, which has progressed to the castration-resistant stage.
2. Ongoing androgen deprivation therapy (ADT) with a gonadotropin-releasing hormone analog or status post bilateral orchiectomy, with serum testosterone < 50 ng/dL (< 1.73 nmol/L) within 28 days prior to study enrollment. Patients receiving ADT at the time of enrollment should continue this therapy throughout the study period.
3. Presence of a predicted loss-of-function BRCA1/2 mutation in germline or tumor tissue.
4. Received at least > 2 lines of systemic therapy for advanced disease (must have received a novel hormonal agent [NHA] and chemotherapy), with recent radiological confirmation of disease progression.

Cohort 4:

1) The aforementioned tumor types (from Cohorts 1-3) harboring HRRm (excluding BRCA mutations), or other tumor types harboring HRRm (including but not limited to esophageal cancer, small cell lung cancer, or pancreatic cancer, etc.), which have failed after first-line or later standard therapy.

3. Presence of at least one measurable lesion according to RECIST v1.1. 4. For both Phase I backfill and Phase II expansion, patients must provide tumor tissue (archived specimen from within 12 months pre-ICF preferred; fresh biopsy if unavailable) and peripheral blood for BRCAm/HRRm testing. Provision of specimens is also encouraged for Phase I dose-escalation patients when feasible. Testing will be conducted at a Sponsor-designated central laboratory. The samples provided shall comply with the following requirements:

* Option 1 : 8-10 sections of surgically resected tumor tissue specimens, or 10-15 sections of core needle biopsy specimens; fine needle aspiration specimens are not acceptable; plus approximately 2 mL of peripheral blood.
* Option 2 : If tumor tissue samples cannot be provided, a peripheral blood sample of approximately 10 mL may be provided instead.

Note:BRCAm/HRRm results must meet eligibility criteria. A prior positive local laboratory report is acceptable for enrollment without awaiting central lab results; the central report will serve for retrospective validation. If sample quantity is insufficient, Sponsor consultation is required for enrollment eligibility.

5. ECOG Performance Status of 0-1. 6. Expected survival time ≥ 3 months. 7. Adequate organ function:

a. Hematopoietic system (Has not received blood transfusion or hematopoietic growth factor therapy within 14 days): i. Platelet count ≥ 100 × 10^9/L ii. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L iii. White blood cell count ≥ 3.0 × 10^9/L iv. Hemoglobin ≥ 90 g/L b. Hepatic function: i. Total bilirubin ≤ 1.5 × ULN ii. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN (in the absence of liver metastases) iii. ALT and AST ≤ 5.0 × ULN (In subjects with liver metastases) c. Renal function: i. Creatinine clearance (Ccr) > 50 mL/min (calculated by the Cockcroft-Gault formula) d. Coagulation function: i. Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN ii. International normalized ratio (INR) ≤ 1.5 × ULN 8. Both PARPi-pretreated and PARPi-naive patients are eligible for enrollment. For PARPi-pretreated patients, they are allowed to have received a maximum of one prior line of PARPi-containing therapy (whether as monotherapy or as maintenance therapy).

9. Women of childbearing potential (WOCBP) (defined as those not surgically sterile or from menarche until 1 year after menopause) must have a negative serum pregnancy test result within 7 days prior to the first dose of the IP. WOCBP must agree to practice abstinence or use highly effective contraceptive methods from the time of signing the informed consent form until 3 months after the last dose of the IP. Similarly, male subjects (including those post-vasectomy) must agree to use effective contraception or practice abstinence from the time of signing the informed consent until 3 months after the last dose of the IP, and must refrain from sperm donation during this period.

10. The subject must provide informed consent for the study prior to any trial-related procedures and voluntarily sign the written informed consent form.

Exclusion Criteria:

1. Have received systemic anti-tumor therapy (including chemotherapy, biotherapy, endocrine therapy, immunotherapy, etc.) within 4 weeks prior to the first dose of the investigational product, with the following specifics: mitomycin and nitrosoureas within 6 weeks from the last dose; oral fluorouracil drugs (such as tegafur and capecitabine) within 2 weeks from the last dose; small molecule targeted agents within 2 weeks or 5 half-lives from the last dose, whichever is shorter; have received any herbal or botanical products with purported anti-tumor effects within 2 weeks prior to the first dose of the investigational product.
2. Have received radiotherapy (with the exception of palliative radiotherapy) within 3 weeks prior to the initiation of study treatment, or have a history of radiation pneumonitis. Note: With the exception of a history of radiation pneumonitis, subjects must have recovered from all radiation-related toxicities.
3. Have received other unapproved investigational drugs within 4 weeks prior to the first dose of the investigational product, or within 5 half-lives of the other drug(s), whichever is shorter.
4. Have undergone major organ surgery (excluding Puncture Biopsy) within 4 weeks prior to the first dose of the investigational product, or have experienced significant trauma, or require elective surgery during the trial period.
5. Prior treatment with a PARP1 inhibitor. Note: For subjects enrolling in the dose-escalation phase, enrollment may be considered following discussion with and agreement from the sponsor's medical representative.
6. Have received or are anticipated to require long-term systemic glucocorticoid therapy (prednisone >10 mg/day or equivalent) or other immunosuppressive therapy within 14 days prior to the first dose of the investigational product. The following are exceptions: topical, intra-articular, intranasal, and inhaled corticosteroids; corticosteroid administration as premedication for contrast-enhanced imaging studies to prevent allergic reactions; short-term (≤ 7 days) use of corticosteroids for the prevention or treatment of non-autoimmune allergic conditions; and glucocorticoids used during the treatment stage for castration-resistant prostate cancer (CRPC).
7. Have used immunomodulatory agents, including but not limited to thymic peptides, interleukin-2 (IL-2), interferon, etc., within 14 days prior to the first dose of the investigational product.
8. Have received a live or attenuated live vaccine within 4 weeks prior to the first dose of the investigational product. Inactivated vaccines are permitted.
9. Have used within 7 days prior to the first dose of the investigational product or require concomitant use during the study treatment period of medications, herbal supplements, or foods known to be strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers (refer to Appendix 4 a summary list of common CYP3A4 enzyme inducers and inhibitors).
10. Have a prior history of allogeneic bone marrow transplantation or solid organ transplantation.
11. Patients with myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or presenting with features suggestive of MDS/AML.
12. Have difficulty swallowing oral medications, or have malabsorption syndrome or any other poorly controlled gastrointestinal disease that may affect bioavailability.
13. Adverse reactions from prior anti-tumor therapy have not recovered to ≤ Grade 1 per CTCAE v5.0 (except for alopecia, hyperpigmentation, and other tolerable events judged by the investigator) or to the level specified in the protocol inclusion/exclusion criteria.
14. Patients with central nervous system (CNS) metastases meeting any of the following criteria: (a) requiring local therapy (surgery, radiotherapy, or other); (b) CNS metastases requiring or currently being treated with corticosteroids at a dose >10 mg prednisone or equivalent; (c) unstable CNS metastases or a stability duration of less than 14 days after the last treatment prior to enrollment; (d) presence of spinal cord compression or leptomeningeal metastasis.
15. Presence of severe chronic or active infection requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days prior to the first dose (including tuberculosis infection).
16. Have a known history of a positive human immunodeficiency virus (HIV) test or acquired immunodeficiency syndrome (AIDS).
17. Patients with active hepatitis B (if hepatitis B surface antigen is positive, HBV-DNA testing is required; subjects with positive HBsAg and HBV-DNA > 500 copies/mL or > 100 IU/mL are considered to have active hepatitis B and must be excluded). Subjects who test positive for HBV-DNA may be enrolled if, after receiving antiviral therapy, their HBV-DNA level decreases to below the lower limit of detection for ≥ 2 weeks, and they must continue to receive antiviral therapy during the study period; patients with hepatitis C (if the HCV antibody test is positive, HCV-RNA testing is required; subjects with a positive HCV antibody test and a positive HCV RNA result are considered to have hepatitis C and must be excluded); patients with active syphilis (if the Treponema pallidum antibody test is positive, an antibody titer test is required; patients with active syphilis should be excluded according to the central laboratory's testing standards).
18. History of other malignancies within the past 3 years, except for adequately treated basal cell carcinoma of the skin, superficial bladder cancer, or carcinoma in situ of the cervix.
19. Have a history of severe cardiovascular or cerebrovascular diseases, including but not limited to:

    1. Severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, second- or third-degree atrioventricular block, QTcF interval ≥ 470 ms, etc.
    2. Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other Grade 3 or higher cardiovascular or cerebrovascular events occurring within 6 months prior to the first dose of the investigational product.
    3. For patients with chronic cardiac disease, New York Heart Association (NYHA) functional class > II or left ventricular ejection fraction (LVEF) < 50%.
    4. Poorly controlled hypertension, defined as systolic blood pressure (SBP) ≥ 160 mmHg and/or diastolic blood pressure (DBP) ≥ 100 mmHg despite clinical therapy.
    5. History of severe hemorrhage or thrombotic diseases within 6 months prior to the investigational product administration, or use of anticoagulants (such as warfarin) or similar agents requiring therapeutic International Normalized Ratio (INR) monitoring.
20. Have clinically significant severe pulmonary impairment, including but not limited to infectious pneumonia or requiring continuous supplemental oxygen to maintain adequate oxygenation.
21. Subjects with active autoimmune disease, or a history of autoimmune disease that may recur (including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vasculitis, psoriasis, autoimmune thyroid disease), or subjects with related risks (e.g., those who have undergone organ transplantation requiring immunosuppressive therapy). Subjects with skin diseases that do not require systemic therapy (e.g., vitiligo, psoriasis) may be enrolled.
22. Known hypersensitivity or allergy to any component of the investigational product.
23. Clinically uncontrolled pericardial effusion, pleural effusion, or ascites requiring repeated drainage.
24. Have dementia or altered mental status that may affect the understanding and provision of informed consent.
25. Pregnant or lactating women.
26. Have underlying disease conditions (including laboratory abnormalities), or alcohol/drug abuse or dependence, which may interfere with the administration of the investigational product, affect the interpretation of drug toxicity or adverse events, or lead to inadequate or reduced compliance with study procedures.
27. Any other significant condition that, in the judgment of the investigator, would substantially increase the risk associated with the patient's participation in the study, or affect the patient's ability to receive the investigational product or complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
DLT/MTD | Within 24 days after the first dose (including 3 days of Cycle 0 and 21 days of Cycle 1)
  Incidence and characteristics of Dose-Limiting Toxicity (DLT) to determine the Maximum Tolerated Dose (MTD).
RP2D | From the first dose until disease progresses or end of treatment for other reasons，up to 1 year
  Recommended Phase II Dose (RP2D) of SPR1020, as the dose for efficacy study in Phase II, will be the dose with promising clinical responses observed in the patients, and well tolerated by patients.
Incidence and characteristics of AEs and SAEs (according to NCI CTCAE 5.0) | All AEs/SAEs (including irAEs/AESIs) will be collected from first dose until 30 days after the last dose, or until new anti-tumor therapy begins，up to 1 year
  Incidence and characteristics of Adverse Events (AEs) and Serious Adverse Events (SAEs) throughout the study period, were evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) V5.0.

SECONDARY OUTCOMES:
ORR | From date of first dose until the date of first documented progression, death from any cause, loss of follow-up, withdrawal of informed consent, or study termination by the sponsor, whichever came first，up to 1 year
  Objective Response Rate (ORR) is the proportion of patients with Complete Response (CR) or Partial Response (PR). ORR and other efficacy evaluation indexes are based on RECIST 1.1 criteria
DCR | From date of first dose until the date of first documented progression, death from any cause, loss of follow-up, withdrawal of informed consent, or study termination by the sponsor, whichever came first，up to 1 year
  Disease control rate (DCR) is the proportion of patients with CR, PR, and Stable Disease (SD).
DOR | From date of first dose until the date of first documented progression, death from any cause, loss of follow-up, withdrawal of informed consent, or study termination by the sponsor, whichever came first，up to 1 year
  Duration of Response (DOR) is the time between the first onset of CR or PR and the first onset of Disease Progression (PD) or death from any cause.
PFS | From date of first dose until the date of first documented progression, death from any cause, loss of follow-up, withdrawal of informed consent, or study termination by the sponsor, whichever came first，up to 1 year
  Progression-Free Survival (PFS) is the time between first initiation of study treatment to PD or death due to any reason.
OS | From date of first dose until the date of first documented progression, death from any cause, loss of follow-up, withdrawal of informed consent, or study termination by the sponsor, whichever came first，up to 1 year
  Overall Survival (OS) is defined as the time interval from the date of the first dose of study drug to the date of death from any cause.
Cmax | Up to approximately 189 days(Cycle 9 Day 1，a cycle for 21 days)
  Peak concentration (Cmax).
Tmax | Up to approximately 189 days(Cycle 9 Day 1，a cycle for 21 days)
  Peak time (Tmax).
t1/2 | Up to approximately 189 days(Cycle 9 Day 1，a cycle for 21 days)
  Elimination phase half-life (t1/2).
AUC0-t | Up to approximately 189 days(Cycle 9 Day 1, a cycle for 21 days)
  Area under plasma concentration-time curve from 0 to the last quantifiable time point (AUC0-t).
AUC0-∞ | Up to approximately 189 days(Cycle 9 Day 1, a cycle for 21 days)
  Area under plasma concentration-time curve from 0 to infinite time (AUC0-∞)
AUC0-last | Up to approximately 189 days(Cycle 9 Day 1, a cycle for 21 days)
  Area Under the Concentration-Time Curve from Time 0 to Last Quantifiable Concentration.
CL | Up to approximately 189 days(Cycle 9 Day 1, a cycle for 21 days )
  Clearance
Vd | Up to approximately 189 days(Cycle 9 Day 1, a cycle for 21 days)
  Volume of Distribution
F | Up to approximately 189 days(Cycle 9 Day 1, a cycle for 21 days)
  Bioavailability
PARylation | Up to approximately 15 Days
  Poly(ADP-ribosyl)ation

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The Affiliated Tumor Hospital of Harbin Medical University, Harbin, Heilongjiang